CLINICAL TRIAL: NCT05384236
Title: A Comparative Study of Kinesiology Taping Versus Taping in the Treatment of Plantar Fasciitis
Acronym: Taping
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, CARMEN GARCÍA GOMARIZ, Principal investigator, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UNIVERSIDAD DE VALENCIA
Record Dates: First submitted 2022-03-24; First posted 2022-05-20 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Plantar Fasciitis
MeSH Terms: conditions — Fasciitis, Plantar

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- kinesiology taping (Experimental): Application of a neuromuscular bandage on the plantar fascia
  Interventions: Other: kinesiology taping
- taping or Low-dye taping (Active Comparator): Application of a taping on the plantar fascia
  Interventions: Other: taping or Low-dye taping

INTERVENTIONS:
Other: kinesiology taping — To apply kinesiology taping in plantar fascia
  Arms: kinesiology taping
Other: taping or Low-dye taping — To apply taping or Low-dye taping in plantar fascia
  Arms: taping or Low-dye taping

SUMMARY:
Plantar fasciitis is a very studied pathology and treated with taping. There are studies that assess the effectiveness of Kinesio taping, as well as taping or low-dye taping, few studies that compare the two treatments and assess which is more effective.

In the present work the effectiveness of Kinesio taping and taping will be assessed, as well as whether possible differences among intervention effects exist in terms of pain improvement, comfort and durability of the bandage.

ELIGIBILITY:
Inclusion Criteria:

* People with plantar fasciitis.
* People of legal age.

Exclusion Criteria:

* Healthy people
* Minors.
* People with pathologies other than plantar fasciitis in the foot.
* People who have treatment for fasciitis at the time of starting the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2022-10-29 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale of Pain | seven days
  It is rated on a scale of 0 to 10, where 0 is no pain and 10 is extreme pain.
comfort | seven days
  Comfort is rated on a scale of 0 to 10, where 0 is no comfotable and 10 is very comfortable
Visual Analogue Scale of Mobility | seven days
  the degree of MOBILITY that the foot has had when using the bandage, rated from 0 no mobility to 10
Visual Analogue Scale of comfort | seven days
  The degree of COMFORT IN HYGIENE of the bandage: (for example at the time of showering or personal hygiene), rated from 0, no comfort to 10, maximum confort

CONTACTS AND LOCATIONS:
Locations (1):
- Universitat de València, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided